CLINICAL TRIAL: NCT02804048
Title: Physiotherapy Intervention in Climacteric Women With Dyspareunia: A Randomized Controlled Trial
Brief Title: Physiotherapy Intervention in Climacteric Women With Dyspareunia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-0307
Record Dates: First submitted 2016-02-12; First posted 2016-06-17 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Dyspareunia
Keywords: Dyspareunia; Pelvic floor muscles; Women
MeSH Terms: conditions — Dyspareunia | interventions — Musculoskeletal Manipulations; Contraceptive Devices, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvic Floor Muscle Training (Experimental): superficial heat pelvic floor muscle intra vaginal manual therapy. PERFECT scale is applied in 5 sessions and based on the result of each assessment is performed the treatment plan with exercises of the pelvic floor muscles.
  It is performed manual therapy in iliopsoas, diaphragm and piriformis. From the fourth session, initiate treatment with electromyographic biofeedback based on the result of PERFECT scale.
  Interventions: Other: superficial heat pelvic floor muscle; Other: Pelvic Floor Muscle Training; Other: Manual therapy in iliopsoas, diaphragm and piriformis; Other: Intra Vaginal Manual therapy; Other: Electromyographic biofeedback
- Low back (Placebo Comparator): superficial heat low back Manual therapy in piriform, lumbar, iliopsoas and diaphragm.
  Interventions: Other: superficial heat low back; Other: Manual therapy in iliopsoas, diaphragm and piriformis

INTERVENTIONS:
Other: superficial heat pelvic floor muscle — Superficial heat application in the pelvic floor muscle
  Arms: Pelvic Floor Muscle Training
Other: superficial heat low back — Superficial heat application in the low back
  Arms: Low back
Other: Pelvic Floor Muscle Training — Pelvic floor muscle training exercises
  Arms: Pelvic Floor Muscle Training
Other: Manual therapy in iliopsoas, diaphragm and piriformis — Manual therapy in iliopsoas, diaphragm and piriformis for 10 minutes
Other: Intra Vaginal Manual therapy — Intra Vaginal Manual therapy in the pelvic floor muscles
  Arms: Pelvic Floor Muscle Training
Other: Electromyographic biofeedback — Electromyographic biofeedback in the pelvic floor muscles
  Arms: Pelvic Floor Muscle Training

SUMMARY:
Aim: To evaluate the effectiveness of physical therapy intervention techniques in the improvement of dyspareunia in climacteric women.

Study design: This is a randomized controlled trial.

DETAILED DESCRIPTION:
Search location: Menopause and Sexuality Clinic of the department of obstetrics and Gynecology and Clinical Research Center, Hospital de Clínicas de Porto Alegre (HCPA).

Patients or participants: The recruited patients may not be vaginal atrophy (cytology-hormone test) and must provide the diagnosis of dyspareunia for more than six months being confirmed by one of the investigators through the pain score above grade 3 (visual analog pain scale) visual inspection, palpation and a questionnaire about the duration and location of pain.

Intervention and measures: consist of evaluation of the pelvic floor muscles (Oxford Scale and Perfect), myoelectric assessment (Electromyography), quality of life (Cervantes Scale), sexual function (FSFI), level of depression (Beck Scale) and pain (visual analog pain scale) before and after physical therapy intervention.

Expected results: To estimate the effectiveness of pelvic floor training techniques with physical therapy in women with dyspareunia.

ELIGIBILITY:
Inclusion Criteria:

* dyspareunia complaint for at least six months
* visual analog scale of pain above 3
* trophic vagina

Exclusion Criteria:

* vaginal atrophy
* neurological disorders
* lack of cognition and understanding
* urinary tract infection and / or genital infections
* prolapse grade 2 and 3
* severe systemic disease
* performing physical therapy

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-12; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of physiotherapy techniques in pain improvement using visual analog scale pain | Seven meetings, twice a week, in which the first is the initial assessment and the seventh is the final evaluation totaling a maximum of one month treatment for each patient.
  To evaluate the effectiveness of physiotherapy techniques using the analog pain scale.

SECONDARY OUTCOMES:
To evaluate the quality of life | To evaluate the quality of life, using Cervantes Scale in climateric women in baseline and after four weeks of intervention
To evaluate depression | To evaluate depression, using Beck Scale, in baseline and after four weeks of intervention
To evaluate sexual function | To evaluate sexual function, using Female Sexual Function Index, in baseline and after four weeks of intervention
To evaluate electrical activity of the pelvic floor muscles | To evaluate electrical activity of the pelvic floor muscles, using Electromyographic biofeedback , in baseline and after four weeks of intervention
To evaluate the pelvic floor muscle function | To evaluate the pelvic floor muscle function, using PERFECT Scale in baseline and after four weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Maria Celeste Wender, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Clinical Research Center of HCPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided